CLINICAL TRIAL: NCT05952349
Title: Effect of Metformin and Combination of Olive Oil Plus Nutritional Supplements on Inflammatory Markers IL-6 and IL-8 in PCOS.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Khyber Medical University Peshawar (Other)
Responsible Party: Principal Investigator, Mohsin Shah, Associate Professor, Khyber Medical University Peshawar
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NO:KMU/IBMS/2023/75
Record Dates: First submitted 2023-07-11; First posted 2023-07-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: PCO
Keywords: Metformin; L-Carnitine; Interleukin-6; L-arginine; CoQ-10
MeSH Terms: interventions — Olive Oil; Metformin

STUDY DESIGN:
Intervention Model Description: cross-sectional study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combination Therapy Group (Active Comparator): ARM# 1 OLIVE OIL 5ML/5MG (BD) NUTRITIONAL SACHET 2100MG (BD)
  Interventions: Drug: OLIVE OIL 5ML/5MG (BD) NUTRITIONAL SACHET 2100MG (BD)
- Standard Therapy Group (Other): ARM # 2 METFORMIN 1000MG (BD)
  Interventions: Drug: Metformin (1000 mg Twice a day)

INTERVENTIONS:
Drug: OLIVE OIL 5ML/5MG (BD) NUTRITIONAL SACHET 2100MG (BD) — 44 Patients with PCOS receiving olive oil 5ML/5MG (BD) nutritional sachet 2100MG (BD
  Arms: Combination Therapy Group
Drug: Metformin (1000 mg Twice a day) — 44 Patients with PCOS receiving Metformin 1000mg (BD)
  Arms: Standard Therapy Group

SUMMARY:
The investigators aim is to conduct randomized clinical trial, to determine the effects of metformin and combination of olive oil plus nutritional supplements on inflammatory markers IL-8 and IL6 in polycystic ovarian syndrome (PCOS). Women diagnosed with PCOS using "Rotterdam diagnostic criteria" according to which two out of three characters must be their in women of PCOS. The investigators propose that PCOS women have increase levels of IL-6 ,IL-8 and this therapy would have beneficial effects and is able to reduce their increase interleukins levels .

DETAILED DESCRIPTION:
Poly cystic ovary syndrome (PCOS) is an endocrine and metabolic disorder, it affects approximately 4% to 7% of women of child bearing age. PCOS is characterized by poly cystic ovaries, an-ovulation, and other associated features of hyperandrogenism It is pro inflammatory state which is related to insulin resistance, irregular menstruation(oligomenorrhea), type II diabetes, hyperinsulinemia and increased hair growth as signs and symptoms An anti-hyperglycemic agent such as Metformin improves glucose tolerance, and at cellular levels increase the action of insulin without affecting it's secretion. Insulin resistance, hyperinsulinemia and lipid abnormalities are managed by treatment with metformin. Several studies indicate a positive effect of metformin on both metabolic and reproductive aspects in female having PCOS. Metformin is known to reduce obesity and decrease other inflammatory biomarkers like serum c-reactive protein in female having PCOS.

L-carnitine is synthesized by the human body as an endogenous compound, it plays a very important role in the metabolism of fatty acid. L-Carnitine is a cofactor and it help in the oxidation of fatty acids by transporting long-chain of fatty acids across mitochondrial membrane. LC levels are found reduced in patients having PCOS; therefore, for the proper management for insulin resistance and obesity in women adjunctive therapy of LC could be beneficial.

Recent studies on olive oil shows that it helps in reducing fatty liver, while olive oil consumption had no effects on the lipid profile. Olive oil has excellent anti-inflammatory potentials against IL-6,IL-8 and TNF produced into the bloodstream as compared to metformin. As a result, it can be used in PCOS treatment.

IL-6 shows an essential part in endocrine system as a major pro-inflammatory cytokine, particularly related to ovarian growth and the course of fertilization and implantation. IL-6 is involved in low grade chronic inflammation in female with PCOS2. IL-6 also showed to have an effect on insulin resistance and cardiovascular abnormalities . Elevated IL-6 levels is reported to be associated with increase weight, a major risk factor for type II diabetes.

IL-8 is proinflammatory cytokine.Il-8 is chemoattractant and it activate neutrophils. Proinflammatory markers like il-6 and il-8 are involved in the development in development of insulin resistance in PCO. Insulin resistance is involved in exaggeration of inflammatory process.

Arginine is amino acid by nature. It is an essential substrate for nitric oxide synthesis which is involved in insulin signaling. Its supplementation can improve metabolic disorders, immune function, wound healing, lean tissue mass, and brown adipose tissue growth.Co-q10 act as a cofactor in the electron transport chain and in the series of redox reaction which are crucial in the synthesis of adenosine tri phosphate. Co-Q10 is essential of the health of almost all organs and tissues because ATP is the soul requirement of all cellular functions. Coq-10 is the most important lipid antioxidants, it guards against the formation of free radicals and their alterations to proteins, lipids, and DNA.

PCOS is an anti-inflammatory condition. Previous studies shows that level of certain cytokines are elevated in individual with PCOS. Studies related to inflammatory markers and PCOS are very few so, this research will help us in better understanding of inflammatory markers and PCOS and it will also help us in deciding a more better treatment plan for female patients having PCOS.The purpose of this study is to determine the effects of metformin and combination of olive oil plus nutritional supplements after 3 months, on inflammatory markers IL-8 and IL6 in polycystic ovarian syndrome

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed according to Rotterdam criteria (2 out of 3 should be present)

  1. Hyperandrogenism
  2. Polycystic ovaries
  3. Menstrual irregularities
* Age 18-34 years

Exclusion Criteria:

* Previous history of Cushing's syndrome
* Women using other medications simultaneously which may affect hormonal changes
* Previous history of ovarian surgery
* Congenital adrenal hyperplasia
* Thyroid diseases
* Autoimmune diseases

  * •

Ages: 18 Years to 34 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Interleukin 6 level | 3 months
  measurement of IL-6 level vis ELISA
Interleukin 8 level | 3 months
  measurement of IL-8 level vis ELISA

CONTACTS AND LOCATIONS:
Overall Officials: Mohsin Shah, PHD, Principal Investigator — Department of Physiology, Khyber Medical University, Peshawar Pakistan
Locations (1):
- Gynecology and Obstetric, Hayatabad Medical Complex, Peshawar, Khyber Pakhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ortega-Gonzalez C, Luna S, Hernandez L, Crespo G, Aguayo P, Arteaga-Troncoso G, Parra A. Responses of serum androgen and insulin resistance to metformin and pioglitazone in obese, insulin-resistant women with polycystic ovary syndrome. J Clin Endocrinol Metab. 2005 Mar;90(3):1360-5. doi: 10.1210/jc.2004-1965. Epub 2004 Dec 14. PMID 15598674
- [Background] Xu X, Du C, Zheng Q, Peng L, Sun Y. Effect of metformin on serum interleukin-6 levels in polycystic ovary syndrome: a systematic review. BMC Womens Health. 2014 Aug 5;14:93. doi: 10.1186/1472-6874-14-93. PMID 25096410
- [Background] Velazquez EM, Mendoza S, Hamer T, Sosa F, Glueck CJ. Metformin therapy in polycystic ovary syndrome reduces hyperinsulinemia, insulin resistance, hyperandrogenemia, and systolic blood pressure, while facilitating normal menses and pregnancy. Metabolism. 1994 May;43(5):647-54. doi: 10.1016/0026-0495(94)90209-7. PMID 8177055
- [Background] Hwang KR, Choi YM, Kim JJ, Chae SJ, Park KE, Jeon HW, Ku SY, Kim SH, Kim JG, Moon SY. Effects of insulin-sensitizing agents and insulin resistance in women with polycystic ovary syndrome. Clin Exp Reprod Med. 2013 Jun;40(2):100-5. doi: 10.5653/cerm.2013.40.2.100. Epub 2013 Jun 30. PMID 23875167
- [Background] Takemura Y, Osuga Y, Yoshino O, Hasegawa A, Hirata T, Hirota Y, Nose E, Morimoto C, Harada M, Koga K, Tajima T, Yano T, Taketani Y. Metformin suppresses interleukin (IL)-1beta-induced IL-8 production, aromatase activation, and proliferation of endometriotic stromal cells. J Clin Endocrinol Metab. 2007 Aug;92(8):3213-8. doi: 10.1210/jc.2006-2486. Epub 2007 May 15. PMID 17504902
- [Background] Sangeeta S. Metformin and pioglitazone in polycystic ovarian syndrome: a comparative study. J Obstet Gynaecol India. 2012 Oct;62(5):551-6. doi: 10.1007/s13224-012-0183-3. Epub 2012 Oct 16. PMID 24082557
- [Background] Yahay M, Heidari Z, Allameh Z, Amani R. The effects of canola and olive oils consumption compared to sunflower oil, on lipid profile and hepatic steatosis in women with polycystic ovarian syndrome: a randomized controlled trial. Lipids Health Dis. 2021 Jan 29;20(1):7. doi: 10.1186/s12944-021-01433-9. PMID 33514384
- [Background] Peng Z, Sun Y, Lv X, Zhang H, Liu C, Dai S. Interleukin-6 Levels in Women with Polycystic Ovary Syndrome: A Systematic Review and Meta-Analysis. PLoS One. 2016 Feb 5;11(2):e0148531. doi: 10.1371/journal.pone.0148531. eCollection 2016. PMID 26849353
- [Background] Abraham Gnanadass S, Divakar Prabhu Y, Valsala Gopalakrishnan A. Association of metabolic and inflammatory markers with polycystic ovarian syndrome (PCOS): an update. Arch Gynecol Obstet. 2021 Mar;303(3):631-643. doi: 10.1007/s00404-020-05951-2. Epub 2021 Jan 13. PMID 33439300
- [Background] Wu G, Meininger CJ, McNeal CJ, Bazer FW, Rhoads JM. Role of L-Arginine in Nitric Oxide Synthesis and Health in Humans. Adv Exp Med Biol. 2021;1332:167-187. doi: 10.1007/978-3-030-74180-8_10. PMID 34251644
- [Background] Saini R. Coenzyme Q10: The essential nutrient. J Pharm Bioallied Sci. 2011 Jul;3(3):466-7. doi: 10.4103/0975-7406.84471. No abstract available. PMID 21966175